CLINICAL TRIAL: NCT01253057
Title: A Research on the Hospital Pollution Control and Hygine Intervention of Chemotherapy Drugs Exposure
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Taipei Medical University WanFang Hospital (Other)
Responsible Party: Ruey-Yu Chen, Taipei Medical University School of Public Health
Other Study IDs: 99061
Record Dates: First submitted 2010-12-01; First posted 2010-12-03 (Estimated); Last update posted 2010-12-03 (Estimated); Status verified 2010-12

CONDITIONS: Sister-chromatic-exchange(SCE); Micronuclei(MN)
Keywords: cleaning staff; antineoplastic agents

STUDY DESIGN:
Observational Model: Case-Control
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Experimental Group
- Control Group

SUMMARY:
Several epidemiological studies found that exposure to antineoplastic agents were associated with some reproductive, carcinogenic effects, higher rates of advance micronuclei (MN), sister-chromatic-exchange (SCE) and spontaneous abortion. Cleaning staff were potentially exposed to these agents while cleaning ward, ward toilet or other area.

One medical center and one area hospitals in Taipei.Surface wipe samples were collected in the cleaning staff work area, such as ward environment and ward toilet. Urine and blood samples of subjects were collected for exposure examinations. Platinum-containing drugs (Cisplatin, Carboplatin, Oxaliplatin) were used as indicator drugs in environmental (surface wipe samples) and biological (urine and blood samples) samples.

A self-administered questionnaire was used to collect demographic data, working practices, medical and contact history, and perceived work-related symptoms of cleaning staff.

The results of this study will be to reduce exposure to cleaning staff.

ELIGIBILITY:
Inclusion Criteria:

* Only included those who signed the consent study

Exclusion Criteria:

* none

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: cleaning staff
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2010-10; Study Completion 2011-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Ruey-Yu Chen, Principal Investigator — Taipei Medical University
Locations (1):
- Taipei Medical University WanFang Hospital, Taipei, Taiwan